CLINICAL TRIAL: NCT06926621
Title: An Open-label Extension Study Evaluating the Long-term Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-670 in Adult Subjects With Myotonic Dystrophy Type I
Brief Title: A Study of Long-term Safety and Efficacy of VX-670 in Participants With Myotonic Dystrophy Type I
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-670-101; 2024-517983-47-00 (Other: EU CT Number)
Record Dates: First submitted 2025-04-10; First posted 2025-04-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Myotonic Dystrophy Type 1 (DM1)
Keywords: DM 1; Myotonic Dystrophy 1; Myotonic Dystrophy Type 1 (DM1); VX-670; Myotonic Dystrophy; DM; Myotonia; Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Vertex; Entrada; PMO; ASO; Myotonic Muscular Dystrophy; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Dystrophies
MeSH Terms: conditions — Myotonic Dystrophy; Myotonia; Myotonic Disorders; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Dystrophies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-670 (Experimental): Participants will receive multiple doses of VX-670.
  Interventions: Drug: VX-670

INTERVENTIONS:
Drug: VX-670 — Solution for intravenous administration.

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability, efficacy and pharmacokinetics of VX-670 in participants with Myotonic Dystrophy Type I (DM1).

ELIGIBILITY:
Key Inclusion Criteria:

• Completed study drug treatment in parent study VX23-670-001 (NCT06185764)

Key Exclusion Criteria:

• History of any illness or any clinical condition as pre-specified in the protocol

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-07-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Week 108

SECONDARY OUTCOMES:
Change From Baseline in Splicing Index in Muscle Biopsy at Week 24 | Baseline and at Week 24
Maximum Observed Concentration (Cmax) of VX-670 and its Active Component in Plasma | From Day 1 up to Week 96
Area Under the Concentration Versus Time Curve (AUC) of VX-670 and its Active Component in Plasma | From Day 1 up to Week 96
Concentration of VX-670 and its Active Component in Muscle | Baseline and at Week 24

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (2):
  - Wesley Research Institute, Auchenflower
  - Neuroscience Clinical Trials Unit, Alfred Brain, Melbourne
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg - Pulmonology, Leuven, Belgium
- Canada (4):
  - Altasciences Montreal, Montreal
  - Montreal Neurological Institute-Hospital, Montreal
  - University of Ottawa, Ottawa
  - Universite Laval - Neurology, Québec
- Hospital Universitario y Politecnico La Fe - Neurology, Valencia, Spain
- United Kingdom (3):
  - Queen Elizabeth University Hospital - Neurology, Glasgow
  - Leonard Wolfson Experimental Neurology Centre CRF, London
  - Royal Hallamshire Hospital - Neurology, Sheffield

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/